CLINICAL TRIAL: NCT02115282
Title: A Randomized Phase III Trial of Endocrine Therapy Plus Entinostat/Placebo in Patients With Hormone Receptor-Positive Advanced Breast Cancer
Brief Title: Exemestane With or Without Entinostat in Treating Patients With Recurrent Hormone Receptor-Positive Breast Cancer That is Locally Advanced or Metastatic
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2014-00746; NCI-2014-00746 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E2112; E2112 (Other: ECOG-ACRIN Cancer Research Group); E2112 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Breast Adenocarcinoma; HER2/Neu Negative; Locally Advanced Breast Carcinoma; Metastatic Breast Carcinoma; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling; entinostat; exemestane; Goserelin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (exemestane, entinostat) (Experimental): Patients receive exemestane PO QD on days 1-28 and entinostat PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI at baseline, at the end of cycle 3, every 3 cycles, at treatment discontinuation, and during follow-up, collection of blood samples at baseline and day 15 of cycle 1, and collection of archived tissue at baseline.
  Pre/perimenopausal female patients and all male patients also receive goserelin acetate SC on day 1.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Entinostat; Drug: Exemestane; Drug: Goserelin; Drug: Goserelin Acetate; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment
- Arm B (exemestane, placebo) (Placebo Comparator): Patients receive exemestane as in Arm A and placebo PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI at baseline, at the end of cycle 3, every 3 cycles, at treatment discontinuation, and during follow-up, collection of blood samples at baseline and day 15 of cycle 1, and collection of archived tissue at baseline.
  Pre/perimenopausal female patients and all male patients also receive goserelin acetate SC on day 1.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Exemestane; Drug: Goserelin; Drug: Goserelin Acetate; Procedure: Magnetic Resonance Imaging; Other: Placebo Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and archived tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS 275; MS-275; MS275; SNDX 275; SNDX-275; SNDX275
  Arms: Arm A (exemestane, entinostat)
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Drug: Goserelin — Given PO
  Other Names: ICI-118630
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Placebo Administration — Given PO
  Arms: Arm B (exemestane, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies exemestane and entinostat to see how well they work compared to exemestane alone in treating patients with hormone receptor-positive breast cancer that has spread to nearby tissue or lymph nodes (locally advanced) or another place in the body (metastatic). Estrogen can cause the growth of breast cancer cells. Endocrine therapy using exemestane may fight breast cancer by lowering the amount of estrogen the body makes. Entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether exemestane is more effective with or without entinostat in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether the addition of entinostat to endocrine therapy (exemestane) improves progression-free survival (PFS) and/or overall survival (OS) in patients with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative locally advanced or metastatic breast cancer who have previously progressed on a non-steroidal aromatase inhibitor (Al).

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of entinostat in combination with exemestane, and to compare the safety profile to that of endocrine therapy with placebo.

II. To evaluate the objective response rate of exemestane in combination with entinostat or placebo.

III. To evaluate whether the efficacy of exemestane with entinostat varies with changes in acetylation status in peripheral blood mononuclear cells (PBMCs).

IV. To evaluate the time to treatment deterioration (as defined by decrease in health-related quality of life [HRQL], progression, death) of exemestane + entinostat versus exemestane + placebo arms.

V. To evaluate the differences in overall health-related quality of life (HRQL) between the exemestane + entinostat versus exemestane + placebo arms.

VI. To evaluate the difference with respect to specific symptoms that are associated with entinostat, i.e., fatigue, nausea, anorexia and diarrhea, between the exemestane + entinostat versus exemestane + placebo arms.

VII. To measure adherence to protocol therapy. VIII. To evaluate the pharmacokinetics of entinostat in patients with advanced breast cancer.

IX. To evaluate what, if any, patient variables alter the pharmacokinetic profile of entinostat in patients with advanced breast cancer.

EXPLORATORY OBJECTIVES:

I. To collect archival tumor samples and germline deoxyribonucleic acid (DNA) to explore other potential biomarkers of therapeutic efficacy.

II. To collect patient ratings of adverse events (AEs) using select patient-reported outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE) items to evaluate the psychometric properties of PRO-CTCAE items and explore the incorporation of PRO-CTCAE items into a phase III double-blind placebo-controlled trial.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive exemestane orally (PO) once daily (QD) on days 1-28 and entinostat PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) at baseline, at the end of cycle 3, every 3 cycles, at treatment discontinuation, and during follow-up, collection of blood samples at baseline and day 15 of cycle 1, and collection of archived tissue at baseline.

ARM B: Patients receive exemestane as in Arm A and placebo PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI at baseline, at the end of cycle 3, every 3 cycles, at treatment discontinuation, and during follow-up, collection of blood samples at baseline and day 15 of cycle 1, and collection of archived tissue at baseline.

In both arms, pre/perimenopausal female patients and all male patients also receive goserelin acetate subcutaneously (SC) on day 1.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Estrogen receptor (ER) and/or progesterone receptor (PR) positive histologically confirmed adenocarcinoma of the breast with staining of >= 1% cells will be considered positive; receptor status may be based on any time during treatment prior to study randomization, and from any site (i.e. primary, recurrent, or metastatic)
* Patients whose tumors have HER2 immunohistochemistry (IHC) 3+, in situ hybridization (ISH) >= 2.0, or average HER2 copy number >= 6.0 signals per cell are not eligible; receptor status may be based on any time during treatment prior to study randomization, and from any site (i.e. primary, recurrent, or metastatic)
* Patients must have measurable or non-measurable stage III/locally advanced or metastatic carcinoma of the breast where local therapy with curative intent is not possible; lesions must be evaluated =< 4 weeks prior to study randomization; diagnostic-quality computed tomography (CT) scans with both oral and intravenous (IV) contrast are the expected radiologic method, unless an alternative is approved

  * NOTE: Where baseline imaging has already been performed =< 6 weeks prior to study randomization, repeat imaging may not be required
  * NOTE: As of October 16, 2016, accrual of new patients having non-measurable disease has stopped; the planned accrual for this target population has been reached
* Pre/peri- and postmenopausal women and all men are eligible for this trial; postmenopausal is defined as:

  * Age >= 55 years and one year or more of amenorrhea
  * Age < 55 years and one year or more of amenorrhea, with estradiol < 20 pg/ml
  * Age < 55 with prior hysterectomy but intact ovaries, with estradiol < 20 pg/ml
  * Prior bilateral oophorectomy

    * NOTE: Women who do not fit the criteria for being postmenopausal as above are deemed pre-or peri-menopausal; pre/perimenopausal women and all men can enroll provided they agree to receive concomitant luteinizing hormone-releasing hormone (LHRH) agonist; pre/perimenopausal women must have commenced treatment with LHRH agonist at least 4 weeks prior to randomization; if patients have received alternative LHRH agonist prior to study entry, they must switch to goserelin for the duration of the trial
* Sexually active males and pre/perimenopausal women must agree to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study and for 3 months after discontinuation of therapy
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study =< 2 weeks prior to randomization

  * A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients must not have known central nervous system metastasis or a history of central nervous system (CNS) metastases; patients with leptomeningeal disease are not eligible
* Patients must be disease-free of prior invasive malignancies for > 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

  * NOTE: If there is a history of prior malignancy, patients must not be receiving other specific treatment for that cancer
* Patients must meet at least one of the following criteria:

  * Disease progression any time after non-steroidal AI use in the advanced disease setting
  * Relapse while on or within =< 12 months of end of adjuvant non-steroidal AI therapy with or without prior endocrine therapy for advanced disease
  * NOTE: In either setting, treatment with any prior endocrine therapy must be completed >= 2 weeks prior to cycle 1 day 1 (C1D1) of study treatment with the exception of exemestane which is permitted in the advanced disease setting within =< 4 weeks immediately prior to C1D1; prior adjuvant exemestane is allowed if the disease free interval is > 12 months from the discontinuation of exemestane; prior faslodex, everolimus, palbociclib or other cyclin-dependent kinase (CDK) inhibitor (e.g. ribociclib, abemaciclib) use are allowed and must have been completed >= 2 weeks prior to C1D1; failure to adhere to this washout guideline will result in a protocol violation
* Patients may have received only one prior chemotherapy regimen for metastatic disease provided treatment was completed >= 3 weeks prior to randomization
* Patients may be treated with bone modifying agents such as bisphosphonates or RANK-ligand agents (e.g. denosumab) per American Society of Clinical Oncology (ASCO) guidelines; whenever possible, patients requiring bone modifying agents should start treatment >= 7 days prior to study therapy and should continue the same agent throughout study unless clinically compelled to change
* Prior radiotherapy must in general have been completed >= 2 weeks prior to randomization and patients must have recovered from the toxicity of the radiation

  * NOTE: Patients may receive concurrent radiation therapy to painful sites of bony disease or areas of impending fracture as long as sites of measurable or non-measurable disease outside the radiation therapy port are available to follow
* Patients must NOT receive concurrent anti-cancer therapy or investigational agent unless specified in protocol
* Patients must NOT be receiving valproic acid, an histone deacetylase (HDAC) inhibitor, and may not have previously received any HDAC inhibitor prior to enrollment (e.g. valproic acid, entinostat, vorinostat) unless discussed with the study chair; patients must not have received prior HDAC therapy for the treatment of their malignancy
* Patients must have no known allergies to exemestane, entinostat, or medications that have a benzamide structure (e.g., tiapride, remoxipride, clebropride)
* Patients must NOT suffer from medical or psychiatric conditions that would interfere with protocol compliance, the ability to provide informed consent, or assessment of response or anticipated toxicities; this includes uncontrolled intercurrent illness including, but not limited to ongoing or active infection
* Patients must have recovered from all clinically relevant adverse events to grade 1 or baseline due to previous agents administered (except alopecia)
* Patients must have adequate hematologic, liver and renal function =< 28 days prior to randomization

  * NOTE: It is preferred that laboratory values for eligibility be assessed after the last dose of prior treatment, especially in cases where most-recent treatment prior to study entry is chemotherapy
* Hemoglobin (HgB) >= 9.0 g/dL (=< 28 days prior to randomization)
* Platelet count >= 100,000/mcL (=< 28 days prior to randomization)
* Absolute neutrophil count >= 1,500/mcL (=< 28 days prior to randomization)
* Creatinine =< 2.0 mg/dL (=< 28 days prior to randomization)
* Total bilirubin < 1.5 x institutional upper limit of normal (=< 3 mg/dL in case of Gilbert's syndrome) (=< 28 days prior to randomization)
* Transaminases (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) =< 2.5 x institutional upper limit normal (=< 28 days prior to randomization)
* Known human immunodeficiency virus (HIV)-positive patients should have a cluster of differentiation (CD)4 count > 250/mm^3
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have a life expectancy >= 12 weeks
* Patients must be able to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2014-03-29 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2026-06-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin M Connolly, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (655):
- United States (654):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Mercy San Juan Medical Center, Carmichael, California
  - Enloe Medical Center, Chico, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Saint Helena Hospital, St. Helena, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - IU Health Central Indiana Cancer Centers-Fishers, Fishers, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Reid Health, Richmond, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Saint Elizabeth Healthcare Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - York Hospital, York Village, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Tech University Health Sciences Center-El Paso, El Paso, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
- University Of Pretoria, Pretoria, South Africa

REFERENCES:
- [Derived] Connolly RM, Zhao F, Miller KD, Lee MJ, Piekarz RL, Smith KL, Brown-Glaberman UA, Winn JS, Faller BA, Onitilo AA, Burkard ME, Budd GT, Levine EG, Royce ME, Kaufman PA, Thomas A, Trepel JB, Wolff AC, Sparano JA. E2112: Randomized Phase III Trial of Endocrine Therapy Plus Entinostat or Placebo in Hormone Receptor-Positive Advanced Breast Cancer. A Trial of the ECOG-ACRIN Cancer Research Group. J Clin Oncol. 2021 Oct 1;39(28):3171-3181. doi: 10.1200/JCO.21.00944. Epub 2021 Aug 6. PMID 34357781
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on March 19, 2014 and terminated on October 17, 2018 with a total accrual of 608 patients.
Groups:
- Arm A (Exemestane, Entinostat): Patients receive exemestane PO QD on days 1-28 and entinostat PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pre/perimenopausal female patients and all male patients also receive goserelin acetate SC on day 1.
  Entinostat: Given PO
  Exemestane: Given PO
  Goserelin Acetate: Given SC
- Arm B (Exemestane, Placebo): Patients receive exemestane as in Arm A and placebo PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pre/perimenopausal female patients and all male patients also receive goserelin acetate SC on day 1.
  Exemestane: Given PO
  Goserelin Acetate: Given SC
  Placebo Administration: Given PO
Period: Overall Study
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Started | 305 | 303
Eligible | 265 | 257
Treated | 296 | 293
Completed (There was no prespecified maximum cycles in the study. Patients were treated until disease progression or intolerability. At the time the primary results were reported, 6 patients were still receiving treatment and they stopped treatment afterwards.) | 0 | 0
Not Completed | 305 | 303
Not completed — Disease progression during treatment | 216 | 229
Not completed — Adverse Event | 49 | 23
Not completed — Death | 1 | 3
Not completed — Alternative therapy | 1 | 1
Not completed — Complicating disease | 0 | 3
Not completed — Withdrawal by Subject | 12 | 10
Not completed — Symptomatic progression/deterioration | 7 | 18
Not completed — Non-compliance | 5 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Study termination (stop treatment due to the release of the results) | 3 | 3
Not completed — Not start protocol therapy | 9 | 10

BASELINE CHARACTERISTICS:
Population: All randomized patients (ie, intent-to-treat patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo) | Total
Number analyzed (Participants) | 305 | 303 | 608
Age, Continuous [Median (Full Range); unit: years] | 63 [31 to 91] | 63 [29 to 90] | 63 [29 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 300 | 602
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 18 | 36
  Not Hispanic or Latino | 284 | 278 | 562
  Unknown or Not Reported | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 42 | 49 | 91
  White | 246 | 244 | 490
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined to be time from randomization to the earliest documented disease progression as defined by the RECIST criteria, new primary breast cancer, or death without progression. Disease assessment was to continue until disease progression, even after non-protocol anti-cancer therapy was started. Cases with incomplete follow up or without adequate disease evaluations were censored at the date last documented to be free of progression, regardless of whether non-protocol anti-cancer therapy was started or not. Disease progression was based on central review, and defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. In addition, the appearance of one or more new lesions was also considered progression. Kaplan-Meier method was used to estimate PFS rate.
Time Frame: Assessed at baseline, then every 12 weeks until treatment discontinuation, then every 3 months within 2 years from study entry, every 6 months between 2-5 years and annually between 6-10 years from study entry, until first disease progression
Population: The first 360 patients randomized to the trial (primary analysis population for the PFS endpoint)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 180 | 180
months | 3.3 [3.1 to 5.3] | 3.1 [3.0 to 3.3]
Statistical Analysis 1: Comparison: Arm A (Exemestane, Entinostat) vs Arm B (Exemestane, Placebo); Test type: Superiority; p = 0.30, Log Rank — The p value was based on stratified log rank test, the threshold for significance was two-sided p value of 0.2%; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.67 to 1.13]

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined to be time from randomization to death from any cause. Cases who were still alive were censored at the date last known alive.
Time Frame: Assessed every 3 months within 2 years from study entry, every 6 months between 2-5 years and annually between 6-10 years from study entry, until death
Population: All randomized patients (ie, intent-to-treat patients, primary analysis population for the OS endpoint)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 305 | 303
months | 23.4 [21.2 to 25.6] | 21.7 [19.3 to 27.1]
Statistical Analysis 1: Comparison: Arm A (Exemestane, Entinostat) vs Arm B (Exemestane, Placebo); Test type: Superiority; p = 0.94, Log Rank — The p value was based on stratified log rank test, stratified on the four randomization factors. The threshold for statistical significance was two-sided p value of 3.7% after taking into account the five interim analyses of OS into account; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.21]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate was defined as number of patients with complete response (CR) or partial response (PR) divided by all randomized patients. Responses were evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline. CR was defined as disappearance of all target and non-target lesions. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameters), and/or persistence of one or more non-target lesion(s).
Time Frame: as for outcome 1
Population: All randomized patients (ie, the intent-to-treat population)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 305 | 303
percentage of participants | 4.6 [2.5 to 7.6] | 4.3 [2.3 to 7.2]

4. Secondary Outcome: Time-to-treatment Deterioration (TTD)
Description: Time-to-treatment deterioration (TTD) was defined as time from randomization to disease progression or death or worsening of symptoms, whichever occurred first. Disease progression was assessed per RECIST v1.1. Symptoms deterioration was measured by 6 items (GP1, GP2, GP4, GF7, B1, P2, scored 0-24) from the 8-item FACT-Breast Symptom Index (FBSI). Symptom deterioration was defined as two consecutive available decreases of at least 3 points from baseline using the 6-item FBSI in this trial, and the second visit time was used as the time of symptom deterioration in this case, unless it was the final score, for which one decrease was sufficient. Kaplan-Meier method was used to estimate the median TTD and TTD rate at a certain time point. Symptoms were assessed every cycle for the first six months after randomization, every two cycles between 6 months and 1 year. It then were assessed based on the same schedule for tumor assessments until disease progression as specified below.
Time Frame: Disease assessed at baseline, then every 12 weeks until treatment discontinuation, then every 3 months within 2 years from study entry, every 6 months between 2-5 years and annually between 6-10 years from study entry, until first disease progression
Population: The first 360 patients randomized to the trial who received at least one dose of protocol therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 175 | 176
months | 2.9 [2.8 to 3.1] | 2.9 [2.8 to 3.0]

5. Secondary Outcome: Lysine Acetylation Change in CD45 Blood Mononuclear Cells Between C1D1 and C1D15 and PFS in Patients on Arm A
Description: Peripheral blood samples (PBMCs) were collected prior to therapy and on Days 8 and 15 of cycle 1, for assessment of lysine acetylation, using an assay developed by the Trepel Laboratory, NCI/NIH. CD45 blood mononuclear cells were measured. Patients with lysine acetylation change of 1.5 folds or higher were compared to patients with lysine acetylation change of less than 1.5 folds.
Time Frame: as for outcome 4
Population: All patients who were randomized to arm A (exemestane +entinostat) and had lysine acetylation test results at both C1D1 and C1D15
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A (Exemestane, Entinostat)- Lysine Acetylation Change>=1.5 Fold; Arm A (Exemestane, Entinostat)- Lysine Acetylation Change<1.5 Fold: Patients receive exemestane PO QD on days 1-28 and entinostat PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pre/perimenopausal female patients and all male patients also receive goserelin acetate SC on day 1.
  Entinostat: Given PO
  Exemestane: Given PO
  Goserelin Acetate: Given SC
Arm/Group | Arm A (Exemestane, Entinostat)- Lysine Acetylation Change>=1.5 Fold | Arm A (Exemestane, Entinostat)- Lysine Acetylation Change<1.5 Fold
Number analyzed (Participants) | 43 | 146
months | 2.8 [2.5 to 5.1] | 2.7 [2.5 to 5.2]

6. Secondary Outcome: Patient-reported Health-related Quality of Life
Description: Health-related quality of life (HRQL) was measured using Functional Assessment of Cancer Therapy - General (FACT-G). The primary endpoint for HRQL was the FACT-G Trial Outcome Index (TOI) which was an aggregate score of 5 items from the FACT-G-Physical subscale (GP2, GP3, GP4, GP6, and GP7) and 6 items from the FACT-G-Functional subscale (GF1, GF2, GF3, GF4, GF6, and GF7). All items were rated on a 5-point Likert scale from 0 to 4. FACT-G TOI subscale score was calculated based on the scoring manual, subscale score ranges from 0 to 44, and higher scores indicate better quality of life. The primary comparison of HRQL between treatment arms was based on the end of cycle 3 assessment.
Time Frame: Assessed at baseline and end of cycle 3
Population: All randomized patients who reported health-related quality of life data at end of cycle 3 assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 203 | 205
units on a scale | 20.5 (5.0) | 20.9 (4.7)

7. Secondary Outcome: Patient-reported Diarrhea
Description: Diarrhea was measured by Functional Assessment of Chronic Illness Therapy for Patients With Diarrhea (FACIT-Diarrhea) subscale form, which had 11 items, all items were rated on a 5-point Likert scale from 0 to 4. FACIT-Diarrhea subscale score was calculated based on the scoring manual, subscale score ranges from 0 to 44, and higher score indicates less diarrhea. The primary comparison of patient-reported diarrhea between treatment arms was based on the end of cycle 3 assessment.
Time Frame: Assessed at baseline and end of cycle 3
Population: All randomized patients who reported FACIT-Diarrhea data at end of cycle 3 assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 208 | 209
units on a scale | 38.8 (7.2) | 41.5 (4.3)

8. Secondary Outcome: Patient-reported Fatigue
Description: Fatigue was measured by PROMIS Fatigue short form, it had 7 items and all items were rated on a 5-point Likert scale from 1 to 5. The PROMIS Fatigue total score and T score were calculated based on the scoring manual. The total score ranges from 7 to 35, the T score ranges from 29.4 to 83.2, higher scores indicate more fatigue. The PROMIS Fatigue T score was used for arm comparison. The primary comparison of patient-reported fatigue between treatment arms was based on the end of cycle 3 assessment.
Time Frame: Assessed at baseline and end of cycle 3
Population: All randomized patients who reported PROMIS fatigue data at end of cycle 3 assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 201 | 207
T-score | 55.5 (8.2) | 54.1 (8.9)

9. Secondary Outcome: Patient-reported Nausea and Anorexia
Description: Nausea and anorexia were measured by The Functional Assessment of Anorexia/Cachexia Treatment (FAACT)-additional concerns, which had 12 items, all items were rated on a 5-point Likert scale from 0 to 4. FAACT-additional concerns subscale score was calculated based on scoring manual. Subscale score ranges from 0 to 48, and higher scores indicate less nausea and anorexia. The primary comparison of patient-reported nausea and anorexia between treatment arms was based on the end of cycle 3 assessment.
Time Frame: Assessed at baseline and end of cycle 3
Population: All randomized patients who reported FAACT nausea and anorexia data at end of cycle 3 assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A (Exemestane, Entinostat) | Arm B (Exemestane, Placebo)
Number analyzed (Participants) | 208 | 203
units on a scale | 35.8 (7.8) | 37.0 (7.9)

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 cycle=28 days) while on treatment and for 30 days after the end of treatment, up to 10 years from study entry
Description: Only patients who received protocol therapy were included in the analysis of adverse events. All randomized patients were included in the analysis of all-cause mortality.
Groups:
- Arm A (Exemestance, Entinostat): Patients receive exemestane PO QD on days 1-28 and entinostat PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pre/perimenopausal female patients and all male patients also receive goserelin acetate SC on day 1.
  Entinostat: Given PO
  Exemestane: Given PO
  Goserelin Acetate: Given SC
- Arm A (Exemestance, Placebo): Patients receive exemestane as in Arm A and placebo PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Pre/perimenopausal female patients and all male patients also receive goserelin acetate SC on day 1.
  Exemestane: Given PO
  Goserelin Acetate: Given SC
  Placebo Administration: Given PO
Arm/Group | Arm A (Exemestance, Entinostat) | Arm A (Exemestance, Placebo)
All-Cause Mortality (participants affected / at risk) | 209/305 | 203/303
Serious Adverse Events (participants affected / at risk) | 151/296 | 47/293
Other Adverse Events (participants affected / at risk) | 280/296 | 228/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Exemestance, Entinostat) (N=296) | Arm A (Exemestance, Placebo) (N=293)
Anemia (Blood and lymphatic system disorders) | 22 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Heart failure (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Edema limbs (General disorders) | 3 | 1
Edema trunk (General disorders) | 1 | 0
Fatigue (General disorders) | 12 | 3
Non-cardiac chest pain (General disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 12 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Bone infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Alkaline phosphatase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 5
Blood bilirubin increased (Investigations) | 3 | 1
GGT increased (Investigations) | 1 | 0
INR increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 10 | 3
Neutrophil count decreased (Investigations) | 58 | 1
Platelet count decreased (Investigations) | 10 | 2
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 18 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 0
Hypokalemia (Metabolism and nutrition disorders) | 7 | 2
Hyponatremia (Metabolism and nutrition disorders) | 8 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 39 | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 5
Thromboembolic event (Vascular disorders) | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Exemestance, Entinostat) (N=296) | Arm A (Exemestance, Placebo) (N=293)
Anemia (Blood and lymphatic system disorders) | 110 | 55
Edema limbs (General disorders) | 54 | 16
Fatigue (General disorders) | 167 | 108
Abdominal pain (Gastrointestinal disorders) | 37 | 21
Constipation (Gastrointestinal disorders) | 36 | 36
Diarrhea (Gastrointestinal disorders) | 106 | 47
Dyspepsia (Gastrointestinal disorders) | 41 | 15
Nausea (Gastrointestinal disorders) | 120 | 76
Vomiting (Gastrointestinal disorders) | 56 | 33
Bruising (Injury, poisoning and procedural complications) | 18 | 3
Alanine aminotransferase increased (Investigations) | 38 | 35
Alkaline phosphatase increased (Investigations) | 85 | 47
Aspartate aminotransferase increased (Investigations) | 56 | 54
Creatinine increased (Investigations) | 33 | 19
Lymphocyte count decreased (Investigations) | 52 | 23
Neutrophil count decreased (Investigations) | 138 | 12
Platelet count decreased (Investigations) | 188 | 19
Weight loss (Investigations) | 29 | 12
White blood cell decreased (Investigations) | 163 | 39
Anorexia (Metabolism and nutrition disorders) | 62 | 30
Hyperglycemia (Metabolism and nutrition disorders) | 29 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 66 | 10
Hypocalcemia (Metabolism and nutrition disorders) | 81 | 14
Hypokalemia (Metabolism and nutrition disorders) | 22 | 11
Hyponatremia (Metabolism and nutrition disorders) | 37 | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 67 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 24
Dizziness (Nervous system disorders) | 21 | 14
Dysgeusia (Nervous system disorders) | 20 | 8
Headache (Nervous system disorders) | 39 | 16
Insomnia (Psychiatric disorders) | 18 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 33 | 19
Hot flashes (Vascular disorders) | 23 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02115282/Prot_SAP_000.pdf